CLINICAL TRIAL: NCT02981472
Title: A Prospective, Randomized, Open Label, Multi-center Study of the Safety and Pharmacokinetics of Apixaban Versus Vitamin K Antagonist or LMWH in Pediatric Subjects With Congenital or Acquired Heart Disease Requiring Chronic Anticoagulation for Thromboembolism Prevention
Brief Title: A Study of the Safety and Pharmacokinetics of Apixaban Versus Vitamin K Antagonist (VKA) or Low Molecular Weight Heparin (LMWH) in Pediatric Subjects With Congenital or Acquired Heart Disease Requiring Anticoagulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pediatric Heart Network (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV185-362; 2016-001247-39 (EudraCT Number)
Record Dates: First submitted 2016-11-18; First posted 2016-12-05 (Estimated); Results first posted 2022-05-18 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — apixaban; acarboxyprothrombin; Warfarin; Heparin, Low-Molecular-Weight; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Apixaban (Experimental)
  Interventions: Drug: Apixaban
- LMWH/VKA (Active Comparator)
  Interventions: Drug: Vitamin K Antagonist (VKA); Drug: Low Molecular Weight Heparin (LMWH)

INTERVENTIONS:
Drug: Apixaban — Specified dose on specified days
  Other Names: Eliquis
  Arms: Apixaban
Drug: Vitamin K Antagonist (VKA) — Specified dose on specified days
  Other Names: Warfarin
  Arms: LMWH/VKA
Drug: Low Molecular Weight Heparin (LMWH) — Specified dose on specified days
  Other Names: Enoxaparin
  Arms: LMWH/VKA

SUMMARY:
To investigate the safety and pharmacokinetics of apixaban in children with congenital or acquired heart disease who have a need for anticoagulation.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Males and Females, 28 days to < 18 years of age, inclusive
* Congenital or acquired heart diseases requiring chronic anticoagulation for thromboprophylaxis (eg, single ventricle physiology including all 3 stages of palliation, dilated cardiomyopathy, Kawasaki disease with coronary aneurysms, and pulmonary hypertension)
* Eligible participants include those who newly start anticoagulants and those who are currently on VKA or LMWH or other anticoagulants for thromboprophylaxis
* Able to tolerate enteral medication [eg, by mouth, nasogastric tube, or gastric tube]
* Participants 28 days to < 3 months must be able to tolerate oral/nasogastric tube (NGT)/gastric tube (GT) feeds for at least 5 days prior to randomization

Exclusion Criteria:

* Recent thromboembolic events less than 6 months prior to enrollment
* Weight < 3 kg
* Use of aggressive life-saving therapies such as ventricular assist devices (VAD) or extracorporeal membrane oxygenation (ECMO) at the time of enrollment
* Artificial heart valves and mechanical heart valves
* Known inherited bleeding disorder or coagulopathy (e.g. hemophilia, von Willebrand disease, etc.)
* Active bleeding at the time of enrollment
* Any major bleeding other than perioperative in the preceding 3 months
* Known intracranial congenital vascular malformation or tumor
* Confirmed diagnosis of a GI ulcer
* Known antiphospholipid syndrome (APS).

Other protocol defined inclusion/exclusion criteria apply

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (46):
- United States (14):
  - Phoenix Children'S Hospital, Phoenix, Arizona
  - University Of California San Diego, La Jolla, California
  - Children'S Hospital Colorado, Aurora, Colorado
  - Childrens Healthcare Of Atlanta, Atlanta, Georgia
  - Local Institution - 0008, Indianapolis, Indiana
  - Local Institution - 0009, Boston, Massachusetts
  - Local Institution - 0013, Ann Arbor, Michigan
  - Childrens Mercy Hospital, Kansas City, Missouri
  - Local Institution - 0006, Cincinnati, Ohio
  - Childrens Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Local Institution - 0012, Charleston, South Carolina
  - Local Institution - 0011, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Local Institution - 0055, Seattle, Washington
- Local Institution, CABA, Buenos Aires, Argentina
- Local Institution - 0030, Parkville, Victoria, Australia
- Local Institution - 0001, Vienna, Austria
- Brazil (5):
  - Local Institution - 0022, Curitiba, Paraná
  - Instituto De Cardiologia Do Rio Grande Do Sul, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0020, Campinas, São Paulo
  - Instituto de Pesquisa PENSI, São Paulo
  - Universidade Federal De Sao Paulo, São Paulo
- Local Institution - 0015, Toronto, Ontario, Canada
- Local Institution - 0031, HUS, Finland
- Germany (3):
  - Local Institution - 0002, Freiburg im Breisgau
  - Local Institution - 0004, Hamburg
  - Local Institution - 0003, München
- Israel (2):
  - Local Institution - 0047, Petah Tikva
  - Local Institution - 0046, Tel Litwinsky
- Italy (3):
  - Local Institution - 0026, Rome, Roma
  - Local Institution - 0028, Bologna
  - Local Institution - 0027, Milan
- Mexico (4):
  - Local Institution - 0044, León, Guanajuato
  - Local Institution - 0018, Mexico City, Mexico City
  - Local Institution - 0019, Mexico City, Mexico City
  - Local Institution - 0016, Mexico City, Mexico City
- Russia (4):
  - Local Institution, Kazan'
  - Local Institution, Kemerovo
  - Local Institution - 0057, Novosibirsk
  - Local Institution - 0062, Yekaterinburg
- Spain (3):
  - Local Institution - 0049, Barcelona
  - Local Institution, Madrid
  - Local Institution - 0048, Madrid
- United Kingdom (3):
  - Local Institution - 0040, Leicester, Leicestershire
  - Local Institution - 0042, Bristol, Somerset
  - Local Institution, Manchester

REFERENCES:
- [Derived] Payne RM, Burns KM, Glatz AC, Male C, Donti A, Brandao LR, Balling G, VanderPluym CJ, Bu'Lock F, Kochilas LK, Stiller B, Cnota JF 2nd, Rahkonen O, Khan A, Adorisio R, Stoica S, May L, Burns JC, Saraiva JFK, McHugh KE, Kim JS, Rubio A, Chia-Vazquez NG, Meador MR, Dyme JL, Reedy AM, Ajavon-Hartmann T, Jarugula P, Carlson-Taneja LE, Mills D, Wheaton O, Monagle P. Apixaban for Prevention of Thromboembolism in Pediatric Heart Disease. J Am Coll Cardiol. 2023 Dec 12;82(24):2296-2309. doi: 10.1016/j.jacc.2023.10.010. PMID 38057072
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 192 participants were randomized and 188 received treatment
Groups:
- Apixaban: Participants receive thromboprophylaxis with open-label apixaban for up to 12 months or until the need for anticoagulant is resolved, whichever occurs first.
  Participants weighing between >/= 3 and < 35 kg will be administered apixaban twice daily (BID) in doses between 0.2mg and 4 mg depending on body weight.
  Children randomized to the apixaban arm of the study weighing >/= 35 kg will be administered apixaban 5 mg twice daily (BID).
- Low Molecular Weight Heparin (LMWH)/Vitamin K Antagonists (VKA): Participants receive thromboprophylaxis with VKA or LMWH for up to 12 months or until the need for anticoagulant is resolved, whichever occurs first.
  Participants who receive LMWH are allowed to switch to VKA at any time during the study; conversely, Participants having difficulty with VKA may switch to LMWH.
Period: Pre-Treatment Period
Arm/Group | Apixaban | Low Molecular Weight Heparin (LMWH)/Vitamin K Antagonists (VKA)
Started | 129 | 63
Completed | 126 | 62
Not Completed | 3 | 1
Not completed — Participant withdrew consent | 2 | 1
Not completed — Participant no longer meets study criteria | 1 | 0
Period: Treatment Period
Arm/Group | Apixaban | Low Molecular Weight Heparin (LMWH)/Vitamin K Antagonists (VKA)
Started | 126 | 62
Completed (completed treatment for up to 12 months or until anticoagulation is no longer needed, whichever is shorter) | 119 | 60
Not Completed | 7 | 2
Not completed — Adverse Event | 6 | 1
Not completed — Participant withdrew consent | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban | Low Molecular Weight Heparin (LMWH)/Vitamin K Antagonists (VKA) | Total
Number analyzed (Participants) | 129 | 63 | 192
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.96 (4.553) | 7.56 (4.408) | 7.83 (4.499)
Age, Customized [Count of Participants; unit: Participants]
  28 DAYS - < 2 YEARS | 8 | 3 | 11
  2 YEARS - < 6 YEARS | 40 | 22 | 62
  6 YEARS - < 12 YEARS | 49 | 23 | 72
  12 YEARS - < 18 YEARS | 32 | 15 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 23 | 90
  Male | 62 | 40 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 14 | 34
  Not Hispanic or Latino | 105 | 47 | 152
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 109 | 51 | 160
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Composite of Adjudicated Major or Clinically Relevant Non-Major (CRNM) Bleeding Events
Description: The number of participants with adjudicated major or CRNM bleeding events per the Perinatal and Paediatric Haemostasis Subcommittee of International Society on Thrombosis and Haemostasis (ISTH) criteria. Events are adjudicated by a blinded, independent events adjudication committee (EAC).
  Major bleeding satisfies one or more of the following criteria: fatal bleeding, clinically overt bleeding associated with a decrease in hemoglobin of at least 20 g/L (i.e., 2 g/dL) in a 24-hour period, bleeding that is retroperitoneal, pulmonary, intracranial, or otherwise involves the CNS, or bleeding that requires surgical intervention in an operating suite, including interventional radiology.
  CRNM bleeding satisfies one or both of the following criteria: overt bleeding for which blood product is administered and not directly attributable to the subject's underlying medical condition or bleeding that requires medical or surgical intervention to restore hemostasis, other than in an operating room.
Time Frame: From first dose to 2 days after last dose (Up to approximately 12 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Low Molecular Weight Heparin (LMWH)/Vitamin K Antagonists (VKA)
Number analyzed (Participants) | 126 | 62
Participants | 1 | 3

2. Secondary Outcome: The Number of Participants With Thrombotic Events and Thromboembolic Event-Related Death
Description: The number of participants with thromboembolic events (intra-cardiac, shunt, inside Fontan pathway, pulmonary embolism (PE), stroke, other arterial or venous thromboembolic events, etc.) and thromboembolic event-related death detected by imaging or clinical diagnosis.
  Death and thromboembolic events are adjudicated by a blinded, independent events adjudication committee (EAC)
Time Frame: From randomization to 2 days after last dose (Up to approximately 12 months)
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Low Molecular Weight Heparin (LMWH)/Vitamin K Antagonists (VKA)
Number analyzed (Participants) | 129 | 63
Participants
  Thromboembolic event | 0 | 0
  Thromboembolic event-related death | 0 | 0

3. Secondary Outcome: The Number of Participants With Adjudicated Major Bleeding
Description: The number of participants with adjudicated major bleeding events per the Perinatal and Paediatric Haemostasis Subcommittee of International Society on Thrombosis and Haemostasis (ISTH) criteria. Major bleeding events are adjudicated by a blinded, independent events adjudication committee (EAC).
  Major bleeding is defined as bleeding that satisfies one or more of the following criteria:
  * fatal bleeding
  * clinically overt bleeding associated with a decrease in hemoglobin of at least 20 g/L (i.e., 2 g/dL) in a 24-hour period
  * bleeding that is retroperitoneal, pulmonary, intracranial, or otherwise involves the CNS
  * bleeding that requires surgical intervention in an operating suite, including interventional radiology
Time Frame: From first dose to 2 days after last dose (Up to approximately 12 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Low Molecular Weight Heparin (LMWH)/Vitamin K Antagonists (VKA)
Number analyzed (Participants) | 126 | 62
Participants | 1 | 1

4. Secondary Outcome: The Number of Participants With Adjudicated CRNM Bleeding
Description: The number of participants with adjudicated clinically relevant non-major (CRNM) bleeding events per the Perinatal and Paediatric Haemostasis Subcommittee of International Society on Thrombosis and Haemostasis (ISTH) criteria. CRNM bleeding events are adjudicated by a blinded, independent events adjudication committee (EAC).
  CRNM bleeding is defined as bleeding that satisfies one or both of the following criteria:
  * overt bleeding for which blood product is administered and not directly attributable to the subject's underlying medical condition
  * bleeding that requires medical or surgical intervention to restore hemostasis, other than in an operating room
Time Frame: From first dose to 2 days after last dose (Up to approximately 12 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Low Molecular Weight Heparin (LMWH)/Vitamin K Antagonists (VKA)
Number analyzed (Participants) | 126 | 62
Participants | 1 | 2

5. Secondary Outcome: The Number of Participants With All Adjudicated Bleeding
Description: The number of participants with all adjudicated bleeding events
Time Frame: From first dose to 2 days after last dose (Up to approximately 12 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Low Molecular Weight Heparin (LMWH)/Vitamin K Antagonists (VKA)
Number analyzed (Participants) | 126 | 62
Participants | 47 | 23

6. Secondary Outcome: The Number of Participants With Drug Discontinuation Due to Adverse Effects, Intolerability, or Bleeding
Description: The number of participants with drug discontinuation due to adverse effects, intolerability, or bleeding.
Time Frame: From first dose to 2 days after last dose (Up to approximately 12 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Low Molecular Weight Heparin (LMWH)/Vitamin K Antagonists (VKA)
Number analyzed (Participants) | 126 | 62
Participants | 7 | 1

7. Secondary Outcome: The Number of Participant Deaths in the Study
Description: The number of participant deaths in the study.
Time Frame: From first dose to 2 days after last dose (Up to approximately 12 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Low Molecular Weight Heparin (LMWH)/Vitamin K Antagonists (VKA)
Number analyzed (Participants) | 126 | 62
Participants | 0 | 0

8. Secondary Outcome: Maximum Observed Concentration (Cmax)
Time Frame: From first dose up to 6 months after first dose
Population: All treated participants in the apixaban arm with available pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Participants Weight Range 6 to < 9 kg: Participants receive thromboprophylaxis with open-label apixaban for up to 12 months or until the need for anticoagulant is resolved, whichever occurs first.
  Participants weighing between 6 to < 9 kg will be administered 1mg apixaban twice daily (BID).
- Participants Weight Range 9 to < 12 kg: Participants receive thromboprophylaxis with open-label apixaban for up to 12 months or until the need for anticoagulant is resolved, whichever occurs first.
  Participants weighing between 9 to < 12 kg will be administered 1.5mg apixaban twice daily (BID).
- Participants Weight Range 12 to < 18 kg: Participants receive thromboprophylaxis with open-label apixaban for up to 12 months or until the need for anticoagulant is resolved, whichever occurs first.
  Participants weighing between 12 to < 18 kg will be administered 2mg apixaban twice daily (BID).
- Participants Weight Range 18 to < 25 kg: Participants receive thromboprophylaxis with open-label apixaban for up to 12 months or until the need for anticoagulant is resolved, whichever occurs first.
  Participants weighing between 18 to < 25 kg will be administered 3mg apixaban twice daily (BID).
- Participants Weight Range 25 to < 35 kg: Participants receive thromboprophylaxis with open-label apixaban for up to 12 months or until the need for anticoagulant is resolved, whichever occurs first.
  Participants weighing between 25 to < 35 kg will be administered 4mg apixaban twice daily (BID).
- Participants Weight Range ≥ 35 kg: Participants receive thromboprophylaxis with open-label apixaban for up to 12 months or until the need for anticoagulant is resolved, whichever occurs first.
  Participants weighing between ≥ 35 kg will be administered 5mg apixaban twice daily (BID).
Arm/Group | Participants Weight Range 6 to < 9 kg | Participants Weight Range 9 to < 12 kg | Participants Weight Range 12 to < 18 kg | Participants Weight Range 18 to < 25 kg | Participants Weight Range 25 to < 35 kg | Participants Weight Range ≥ 35 kg
Number analyzed (Participants) | 6 | 2 | 28 | 29 | 24 | 35
ng/mL | 185 (48.8) | 218 (23.4) | 222 (39.6) | 244 (30.7) | 249 (37.7) | 203 (35.9)

9. Secondary Outcome: Trough Observed Concentration (Cmin)
Time Frame: From first dose up to 6 months after first dose
Population: All treated participants in the apixaban arm with available pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Participants Weight Range 6 to < 9 kg | Participants Weight Range 9 to < 12 kg | Participants Weight Range 12 to < 18 kg | Participants Weight Range 18 to < 25 kg | Participants Weight Range 25 to < 35 kg | Participants Weight Range ≥ 35 kg
Number analyzed (Participants) | 6 | 2 | 28 | 29 | 24 | 35
ng/mL | 57.9 (90.3) | 82.7 (21.5) | 64.3 (69.5) | 67.4 (58.9) | 73.1 (64.7) | 72.7 (46.8)

10. Secondary Outcome: Area Under the Concentration-Time Curve in One Dosing Interval (AUC (TAU))
Time Frame: From first dose up to 6 months after first dose
Population: All treated participants in the apixaban arm with available pharmacokinetic data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng • h/mL
Arm/Group | Participants Weight Range 6 to < 9 kg | Participants Weight Range 9 to < 12 kg | Participants Weight Range 12 to < 18 kg | Participants Weight Range 18 to < 25 kg | Participants Weight Range 25 to < 35 kg | Participants Weight Range ≥ 35 kg
Number analyzed (Participants) | 6 | 2 | 28 | 29 | 24 | 35
ng • h/mL | 1460 (61.2) | 1840 (20.7) | 1610 (49.6) | 1760 (38.3) | 1840 (43.3) | 1630 (37.3)

11. Secondary Outcome: Time of Maximum Observed Concentration (Tmax)
Time Frame: From first dose up to 6 months after first dose
Population: All treated participants in the apixaban arm with available pharmacokinetic data
Measure: Median (Full Range); unit: hours
Arm/Group | Participants Weight Range 6 to < 9 kg | Participants Weight Range 9 to < 12 kg | Participants Weight Range 12 to < 18 kg | Participants Weight Range 18 to < 25 kg | Participants Weight Range 25 to < 35 kg | Participants Weight Range ≥ 35 kg
Number analyzed (Participants) | 6 | 2 | 28 | 29 | 24 | 35
hours | 2.24 [1.41 to 2.83] | 2.47 [2.23 to 2.71] | 1.72 [0.938 to 3.35] | 1.74 [0.775 to 2.18] | 1.65 [1.26 to 2.85] | 1.85 [1.47 to 2.93]

12. Secondary Outcome: Anti-FXa Activity
Description: Anti-FXa Activity was measured to assess participant plasma apixaban levels.
  125 participants received at least one dose of apixaban and had anti-FXa samples collected that contributed measurements to at least one of the timepoints below.
Time Frame: From first dose up to 6 months after first dose
Population: All treated participants in the apixaban arm that have anti-FXa samples collected
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Apixaban
Number analyzed (Participants) | 125
ng/mL
  Day 1 (4 HRS POSTDOSE): number analyzed (Participants) | 116
  Day 1 (4 HRS POSTDOSE) | 147.69 (7.243)
  Week 2 (PREDOSE): number analyzed (Participants) | 113
  Week 2 (PREDOSE) | 86.24 (7.652)
  Week 2 (2 HRS POSTDOSE): number analyzed (Participants) | 44
  Week 2 (2 HRS POSTDOSE) | 242.34 (18.966)
  Month 3 (2 HRS POSTDOSE): number analyzed (Participants) | 68
  Month 3 (2 HRS POSTDOSE) | 228.88 (14.263)
  Month 6 (PREDOSE): number analyzed (Participants) | 100
  Month 6 (PREDOSE) | 66.93 (6.532)

13. Secondary Outcome: Chromogenic FX Assay (Apparent FX Level)
Description: Chromogenic FX was measured to assess (apparent) FX levels in participants and inhibition of FXa by apixaban.
  125 participants received at least one dose of apixaban and had chromogenic FX assay samples collected that contributed measurements to at least one of the timepoints below.
Time Frame: From first dose up to 6 months after first dose
Population: All treated participants in the apixaban arm that have have chromogenic FX assay samples collected
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Apixaban
Number analyzed (Participants) | 125
Percent
  Day 1 (PREDOSE): number analyzed (Participants) | 115
  Day 1 (PREDOSE) | 58.87 (2.368)
  Day 1 (4 HRS POSTDOSE): number analyzed (Participants) | 117
  Day 1 (4 HRS POSTDOSE) | 18.90 (1.205)
  Week 2 (PREDOSE): number analyzed (Participants) | 52
  Week 2 (PREDOSE) | 35.88 (1.973)
  Week 2 (2 HRS POSTDOSE): number analyzed (Participants) | 45
  Week 2 (2 HRS POSTDOSE) | 21.26 (1.680)
  Month 3 (2 HRS POSTDOSE): number analyzed (Participants) | 67
  Month 3 (2 HRS POSTDOSE) | 18.25 (0.970)
  Month 6 (PREDOSE): number analyzed (Participants) | 69
  Month 6 (PREDOSE) | 36.57 (1.943)

14. Secondary Outcome: The Child and Parent Reports of Pediatric Quality of Life Inventory (PedsQL)
Description: Subjects' quality of life was measured using the PedsQL instrument administered only to English-speaking children/parents. Only subjects who completed the questionnaires at both baseline and post-baseline visits were included in the analyses.
  PedsQL consists of 23 items scored on a 5-point Likert scale from 0 (never) to 4 (almost always) or for the child report for younger children ages 5-7, a 3-point Likert scale: 0 (Not at all), 2 (Sometimes), and 4 (A lot).
  Scores are reverse scored and transformed to a 0-100 scale as follows: 0=100, 1=75, 3=25, 4=0. Higher scores indicate a better HRQOL and/or lower problems.
Time Frame: from randomization up to 12 months after randomization
Population: All randomized English speaking participants 2 years and older with both baseline and post baseline questionnaire scores
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Apixaban | Low Molecular Weight Heparin (LMWH)/Vitamin K Antagonists (VKA)
Number analyzed (Participants) | 129 | 63
Score on a scale
  GENERAL-SPECIFIC MODULE ASSESSED BY CHILD - BASELINE: number analyzed (Participants) | 32 | 18
  GENERAL-SPECIFIC MODULE ASSESSED BY CHILD - BASELINE | 69.64 (15.512) | 60.71 (17.374)
  GENERAL-SPECIFIC MODULE ASSESSED BY CHILD - MONTH 12: number analyzed (Participants) | 32 | 18
  GENERAL-SPECIFIC MODULE ASSESSED BY CHILD - MONTH 12 | 73.37 (19.998) | 64.81 (22.327)
  GENERAL-SPECIFIC MODULE ASSESSED BY PARENT - BASELINE: number analyzed (Participants) | 43 | 25
  GENERAL-SPECIFIC MODULE ASSESSED BY PARENT - BASELINE | 65.61 (16.625) | 65.42 (18.000)
  GENERAL-SPECIFIC MODULE ASSESSED BY PARENT - MONTH 12: number analyzed (Participants) | 43 | 25
  GENERAL-SPECIFIC MODULE ASSESSED BY PARENT - MONTH 12 | 70.00 (19.560) | 70.32 (21.949)
  HEART PROBLEMS AND TREATMENT ASSESSED BY CHILD - BASELINE: number analyzed (Participants) | 34 | 17
  HEART PROBLEMS AND TREATMENT ASSESSED BY CHILD - BASELINE | 65.34 (22.130) | 64.70 (18.465)
  HEART PROBLEMS AND TREATMENT ASSESSED BY CHILD - MONTH 12: number analyzed (Participants) | 34 | 17
  HEART PROBLEMS AND TREATMENT ASSESSED BY CHILD - MONTH 12 | 69.46 (21.119) | 63.44 (19.836)
  TREATMENT II ASSESSED BY CHILD - BASELINE: number analyzed (Participants) | 32 | 17
  TREATMENT II ASSESSED BY CHILD - BASELINE | 87.39 (22.994) | 85.68 (15.857)
  TREATMENT II ASSESSED BY CHILD - MONTH 12: number analyzed (Participants) | 32 | 17
  TREATMENT II ASSESSED BY CHILD - MONTH 12 | 91.77 (10.896) | 86.27 (16.400)
  PERCEIVED PHYSICAL APPEARANCE ASSESSED BY CHILD - BASELINE: number analyzed (Participants) | 33 | 17
  PERCEIVED PHYSICAL APPEARANCE ASSESSED BY CHILD - BASELINE | 75.51 (27.477) | 78.44 (23.390)
  PERCEIVED PHYSICAL APPEARANCE ASSESSED BY CHILD - MONTH 12: number analyzed (Participants) | 33 | 17
  PERCEIVED PHYSICAL APPEARANCE ASSESSED BY CHILD - MONTH 12 | 80.56 (22.408) | 81.37 (30.689)
  TREATMENT ANXIETY ASSESSED BY CHILD - BASELINE: number analyzed (Participants) | 34 | 17
  TREATMENT ANXIETY ASSESSED BY CHILD - BASELINE | 80.52 (23.420) | 60.31 (34.162)
  TREATMENT ANXIETY ASSESSED BY CHILD - MONTH 12: number analyzed (Participants) | 34 | 17
  TREATMENT ANXIETY ASSESSED BY CHILD - MONTH 12 | 80.71 (25.480) | 60.31 (38.333)
  COGNITIVE PROBLEMS ASSESSED BY CHILD - BASELINE: number analyzed (Participants) | 34 | 17
  COGNITIVE PROBLEMS ASSESSED BY CHILD - BASELINE | 69.85 (20.871) | 53.24 (20.382)
  COGNITIVE PROBLEMS ASSESSED BY CHILD - MONTH 12: number analyzed (Participants) | 34 | 17
  COGNITIVE PROBLEMS ASSESSED BY CHILD - MONTH 12 | 68.24 (24.367) | 53.53 (26.796)
  COMMUNICATION ASSESSED BY CHILD - BASELINE: number analyzed (Participants) | 32 | 16
  COMMUNICATION ASSESSED BY CHILD - BASELINE | 66.15 (30.000) | 63.55 (28.998)
  COMMUNICATION ASSESSED BY CHILD - MONTH 12: number analyzed (Participants) | 32 | 16
  COMMUNICATION ASSESSED BY CHILD - MONTH 12 | 70.31 (26.681) | 57.28 (38.948)
  HEART PROBLEMS AND TREATMENT ASSESSED BY PARENT - BASELINE: number analyzed (Participants) | 41 | 25
  HEART PROBLEMS AND TREATMENT ASSESSED BY PARENT - BASELINE | 63.68 (20.727) | 67.71 (22.668)
  HEART PROBLEMS AND TREATMENT ASSESSED BY PARENT - MONTH 12: number analyzed (Participants) | 41 | 25
  HEART PROBLEMS AND TREATMENT ASSESSED BY PARENT - MONTH 12 | 66.37 (20.811) | 69.00 (23.688)
  TREATMENT II ASSESSED BY PARENT - BASELINE: number analyzed (Participants) | 39 | 25
  TREATMENT II ASSESSED BY PARENT - BASELINE | 91.41 (11.557) | 85.27 (17.325)
  TREATMENT II ASSESSED BY PARENT - MONTH 12: number analyzed (Participants) | 39 | 25
  TREATMENT II ASSESSED BY PARENT - MONTH 12 | 90.30 (12.381) | 83.80 (18.915)
  PERCEIVED PHYSICAL APPEARANCE ASSESSED BY PARENT - BASELINE: number analyzed (Participants) | 40 | 25
  PERCEIVED PHYSICAL APPEARANCE ASSESSED BY PARENT - BASELINE | 79.16 (22.571) | 79.66 (22.958)
  PERCEIVED PHYSICAL APPEARANCE ASSESSED BY PARENT - MONTH 12: number analyzed (Participants) | 40 | 25
  PERCEIVED PHYSICAL APPEARANCE ASSESSED BY PARENT - MONTH 12 | 79.38 (21.012) | 74.33 (26.998)
  TREATMENT ANXIETY ASSESSED BY PARENT - BASELINE: number analyzed (Participants) | 41 | 25
  TREATMENT ANXIETY ASSESSED BY PARENT - BASELINE | 61.44 (30.804) | 56.27 (33.997)
  TREATMENT ANXIETY ASSESSED BY PARENT - MONTH 12: number analyzed (Participants) | 41 | 25
  TREATMENT ANXIETY ASSESSED BY PARENT - MONTH 12 | 64.03 (29.567) | 57.77 (34.199)
  COGNITIVE PROBLEMS ASSESSED BY PARENT - BASELINE: number analyzed (Participants) | 41 | 25
  COGNITIVE PROBLEMS ASSESSED BY PARENT - BASELINE | 60.29 (29.558) | 61.60 (25.807)
  COGNITIVE PROBLEMS ASSESSED BY PARENT - MONTH 12: number analyzed (Participants) | 41 | 25
  COGNITIVE PROBLEMS ASSESSED BY PARENT - MONTH 12 | 58.69 (29.560) | 58.53 (33.432)
  COMMUNICATION ASSESSED BY PARENT - BASELINE: number analyzed (Participants) | 38 | 25
  COMMUNICATION ASSESSED BY PARENT - BASELINE | 65.57 (27.342) | 67.33 (28.257)
  COMMUNICATION ASSESSED BY PARENT - MONTH 12: number analyzed (Participants) | 38 | 25
  COMMUNICATION ASSESSED BY PARENT - MONTH 12 | 68.20 (24.037) | 66.17 (28.067)

15. Secondary Outcome: Kids Informed Decrease Complications Learning on Thrombosis (KIDCLOT) IMPACT Score
Description: Subjects' quality of life was measured using the KIDCLOT instrument administered only to English-speaking children/parents. Only subjects who completed the questionnaires at both baseline and post-baseline visits were included in the analyses.
  KIDCLOT Parent inventory uses a 5 point Likert scale from 1 (N/A), 2 (Never), 3 (Rarely), 4 ( Now and then), 5 (Often). Child inventory uses a 4 point Likert scale 1 (N/A), 2 (Never), 3 (Now and then), 5 (Always). Values are scores as follows 1=0, 2=1, 3=2, 4=3, 5=4. Score interpretation is 0 to 100 percent IMPACT of anticoagulation on a child's life therefore, higher scores indicates a more negative effect.
Time Frame: from randomization up to 12 months after randomization
Population: All randomized English speaking participants 6 years and older taking apixaban or warfarin with both baseline and post baseline questionnaire scores. Parent inventory includes only participants age >= 34 weeks old.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Apixaban | Low Molecular Weight Heparin (LMWH)/Vitamin K Antagonists (VKA)
Number analyzed (Participants) | 46 | 30
Score on a scale
  BASELINE CHILD REPORTED - 6 MONTHS: number analyzed (Participants) | 24 | 15
  BASELINE CHILD REPORTED - 6 MONTHS | 24.35 (12.887) | 26.45 (12.114)
  POST BASELINE CHILD REPORTED - 6 MONTHS: number analyzed (Participants) | 24 | 15
  POST BASELINE CHILD REPORTED - 6 MONTHS | 22.81 (13.380) | 22.57 (16.049)
  BASELINE CHILD REPORTED - 12 MONTHS: number analyzed (Participants) | 25 | 14
  BASELINE CHILD REPORTED - 12 MONTHS | 22.50 (11.787) | 25.32 (11.719)
  POST BASELINE CHILD REPORTED - 12 MONTHS: number analyzed (Participants) | 25 | 14
  POST BASELINE CHILD REPORTED - 12 MONTHS | 21.52 (13.251) | 18.01 (10.408)
  BASELINE PARENT REPORTED - 6 MONTHS | 37.97 (20.493) | 39.02 (17.932)
  POST BASELINE PARENT REPORTED - 6 MONTHS | 32.32 (17.060) | 37.94 (20.626)
  BASELINE PARENT REPORTED - 12 MONTHS: number analyzed (Participants) | 43 | 25
  BASELINE PARENT REPORTED - 12 MONTHS | 38.37 (18.874) | 39.36 (16.057)
  POST BASELINE PARENT REPORTED - 12 MONTHS: number analyzed (Participants) | 43 | 25
  POST BASELINE PARENT REPORTED - 12 MONTHS | 31.10 (16.021) | 33.61 (17.943)

ADVERSE EVENTS:
Time Frame: AEs are collected from the first dose date until the last dose date + 2 days/ SAEs are collected from the first dose date until the last dose date + 30 days (Up to approximately 13 months) Participants were assessed for All Cause Mortality from their first dose until the study was completed (up to approximately 57 months)
Arm/Group | Apixaban | Low Molecular Weight Heparin (LMWH)/Vitamin K Antagonists (VKA)
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/62
Serious Adverse Events (participants affected / at risk) | 26/126 | 13/62
Other Adverse Events (participants affected / at risk) | 68/126 | 36/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban (N=126) | Low Molecular Weight Heparin (LMWH)/Vitamin K Antagonists (VKA) (N=62)
Arrhythmia (Cardiac disorders) | 1 | 1
Atrial septal defect acquired (Cardiac disorders) | 0 | 1
Cardiac dysfunction (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 1
Hypoplastic left heart syndrome (Congenital, familial and genetic disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Protein-losing gastroenteropathy (Gastrointestinal disorders) | 1 | 1
Generalised oedema (General disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 1
Dengue fever (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Shunt thrombosis (Injury, poisoning and procedural complications) | 2 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Intracardiac pressure increased (Investigations) | 0 | 1
Pulmonary arterial pressure increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Penile haematoma (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban (N=126) | Low Molecular Weight Heparin (LMWH)/Vitamin K Antagonists (VKA) (N=62)
Diarrhoea (Gastrointestinal disorders) | 12 | 4
Vomiting (Gastrointestinal disorders) | 20 | 9
Pyrexia (General disorders) | 20 | 8
Gastroenteritis (Infections and infestations) | 7 | 4
Nasopharyngitis (Infections and infestations) | 13 | 8
Upper respiratory tract infection (Infections and infestations) | 14 | 4
Contusion (Injury, poisoning and procedural complications) | 9 | 5
International normalised ratio increased (Investigations) | 0 | 4
Dizziness (Nervous system disorders) | 4 | 4
Headache (Nervous system disorders) | 19 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 | 6
Haematoma (Vascular disorders) | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/72/NCT02981472/Prot_SAP_000.pdf